CLINICAL TRIAL: NCT05320770
Title: Role Of Ultrasonography Compared To MR Imaging In Assessment Of Tempromandibular Joint Disorders
Brief Title: Role of Ultrasonography in Assessment of Tempromanbular Joint Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alyaa Mohammed Awad, Resident in Interventional and Diagnostic Department ,Sohag University Hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-02-05
Record Dates: First submitted 2022-02-13; First posted 2022-04-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: TMJ Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMD patients with joint hyper mobility (Experimental)
  Interventions: Procedure: US guided TMJ intra articular injection

INTERVENTIONS:
Procedure: US guided TMJ intra articular injection — therapeutic TMJ intra articulatr injection of blood under sonography guidance to reduce joint hyper mobility

SUMMARY:
Evaluation of US efficiency in assessment of the tempromandibular joint disorders in comparison with MRI as the gold standard for technique validation and evaluation of efficiency of therapeutic intra articular injection under sonographic guidance .

DETAILED DESCRIPTION:
Temporomandibular joint disorders is a common condition, Intra-articular causes of TMD include internal joint derangement, osteoarthritis, capsular inflammation, hypermobility and traumatic injury. The most frequent cause of TMJ dysfunction is internal derangement which refers to an alteration in the normal pathways of motion of the TMJ that largely involves the function of the articular disc, therefore, these alterations have been also referred to as disc derangement , signs of which appear in up to 60-70% of the population. The peak incidence is seen in adults aged 20-40 years. Women are at least four times as likely to suffer from the disorder .

Magnetic resonance imaging (MRI) has provided a noninvasive accurate method of assessing the TMJ without associated radiation risks ,its ability to directly visualize the disc and accurately determine the position of the disc with respect to the condyle of the mandible and eminence of the temporal bone. The examination, however, takes 20 to 45 minutes on average to perform depending on the scanner and protocol, and patients have difficulty keeping still and having their mouths open for extended periods of time, especially if they are experiencing pain. In addition, the examination is costly and access is still limited in many centers. Many patients also experience claustrophobia and are unable to complete or even undergo the examination .

Ultrasound is relatively inexpensive, is readily accessible, and can be performed in most outpatient facilities; studies take only an average of 10 to 15 minutes in total, and it is without any known risks. In addition, US provides the opportunity to converse with patients and identify the exact locations of pain, while the probe can be used as a palpable tool for real-time identification of crepitus, clicking, motion, and snapping sensations.

The following US applications were described: Joint effusion, Internal derangement and disc displacement, mainly anterior with and without reduction, Joint function basing on condylar translation range, TMJ dislocation, Guidance in fine-needle aspiration cytology (FNAC), Guidance for TMJ arthrocentesis and Guidance in TMJ injections, e.g., with steroids , Blood .

ELIGIBILITY:
Inclusion Criteria:

* Male and female diagnosed as TMJ disorders (clinically through history of the presentation and physical examination (site, onset, character of pain, radiation, duration and associated symptoms. This pain may refer to the scalp or neck, and is often exacerbated by mastication, yawning or talking for extended periods. Difficulty opening the mouth, clicking, popping or crepitus within the TMJ itself and brief locking of the mandible on jaw opening and closure and Headache, particularly tension type headache).

Exclusion Criteria:

* Uncooperative patients, systemic disease with TMJ involvement as Rheumatoid, psoriatic, and juvenile idiopathic arthritis. Contraindications for MRI : claustrophobia , metallic implants , pacemaker and prosthetic heart valves .Contraindication for intra articular injection : the patients with bleeding disorders , pregnancy , bony pathology of TMJ , allergy to local anesthetic and those on narcotics or anti depressant .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change of temporomandibular joint imaging by ultrasonography and magnetic resonance imaging . | Ultrasonography at baseline visit and MRI one week after baseline visit .
  Imaging of the temporomandibular joint by ultrasonography and imaging by magnetic resonance imaging .
Change of mobility of the temporomandibular joint before and after ultrasonography guided blood injection . | Baseline visit and three months after the baseline intervention .
  Measuring the temporomandibular joint mobility in millimeters by ultrasonography before and after sonar guided injection .